CLINICAL TRIAL: NCT01805427
Title: Extreme Weights and Antiretroviral Therapy Individual Concentrations
Brief Title: Antiretroviral Therapy and Extreme Weight
Acronym: EXTATIC
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Stephane Mouly, MD PhD, MD PhD, Hopital Lariboisière
Other Study IDs: EXTATIC; EXTATIC (Other: URT)
Record Dates: First submitted 2013-02-28; First posted 2013-03-06 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infection
Keywords: trough concentration; weight; HIV; virological failure
MeSH Terms: conditions — HIV Infections; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients treated with efavirenz: HIV-infected on stable HAART regimen with efavirenz
- patients treated with atazanavir: HIV-infected patients on stable HAART regimen with atazanavir
- patients treated with darunavir: HIV-infected patients on stable HAART regimen with darunavir

SUMMARY:
The concentration of the third agent in antiretroviral therapy [Non Nucleoside Reverse Transcriptase Inhibitor (NNRTI), or boosted Protease inhibitor (PI) ] is different according to the body weight or body composition and therapeutic monitoring may be necessary in overweight HIV patients.

The investigators aim at measuring the individual trough concentrations of interest [at steady state for NNRTI and boosted PI] in overweight and normal weight HIV+ patients.

DETAILED DESCRIPTION:
Our primary endpoint is the individual trough concentrations of interest at steady state for NNRTI or boosted PI; Principal outcome measure: comparison of the concentrations between patients <25kg/m2 and patients<25kg/m2

Secondary endpoints:

* Occurrence of virologic failure
* Occurrence of clinical/biological adverse events
* Percentage of patients with concentration within the therapeutic range
* Body composition Secondary outcome measures: comparison of the occurrence of virologic failure, occurrence or adverse event, patients with concentration within the therapeutic range between groups. Correlation between body composition and concentration.

Methodology, study design:

open-labelled monocentric study.

Sample size:

It will be a descriptive experimental study involving 120 overweight subjects, 120 normal weight subjects

Inclusion criteria :

* Patients with HIV+
* Patients aged more than 18 years old.
* Patient giving its well-informed and free consent.

Study design :

Plasma concentration was performed during the usual clinical follow-up. Study duration: 12 months Duration for a patient: 1 day Investigating center and participating units: one center enrolling the patients and the lab performing drug dosages.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HIV+ receiving one of the following third agent their HAART: efavirenz, atazanavir , or darunavir
* Patients aged > 18 years old.
* Patient giving its well-informed and free consent. Patient giving its well-informed and free consent.

Patients living in France during the study.

Exclusion Criteria:

Treatment with rifampin/rifabutin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients aged 18 years and older, treated with either efavirenz, atazanavir, or darunavir for at least 4 weeks and under stable treatment regimen
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
comparison of the trough concentrations between patients with Body Mass Index (BMI)<25 kg/m2 and patients with BMI >25 kg/m2 | the day of enrollment

SECONDARY OUTCOMES:
comparison of the occurrence of virologic failure within each patient group | the day of enrollment

OTHER OUTCOMES:
occurrence of adverse events in each patient group | the day of enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Lariboisiere, Paris, Île-de-France Region, France